CLINICAL TRIAL: NCT07061353
Title: Effect of Therapeutic Touch on Perceived Stress and Comfort Levels in Hemodialysis Patients: A Randomized Controlled Trial
Brief Title: Effect of Therapeutic Touch on Perceived Stress and Comfort Levels in Hemodialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/08-02
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Therapeutic Touch; Hemodialysis Patients
Keywords: Therapeutic touch; Hemodialysis Patient; Stress; Comfort; Nursing
MeSH Terms: interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The person performing the analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Touch (Experimental): Therapeutic Touch group
  Interventions: Behavioral: Therapeutic touch
- Control (No Intervention): No therapeutic touch group

INTERVENTIONS:
Behavioral: Therapeutic touch — Therapeutic touch will be performed
  Arms: Therapeutic Touch

SUMMARY:
Hemodialysis is a treatment method used in the treatment of acute or chronic renal failure, the main function of which is based on the cleaning of accumulated waste materials in the blood, and is rapidly developing and spreading in parallel with today's technology. Patients undergoing hemodialysis treatment are trying to cope with social and physical problems that may develop due to chronic disease. At the same time, their quality of life is affected due to the psychosocial, economic problems and complications brought about by machine dependency. From past to present, individuals have used various methods to protect/improve their health. Today, in addition to modern medicine, complementary/alternative therapies are increasingly used. One of these alternative therapies is the therapeutic touch application, which has recently gained popularity. Therapeutic touch is based on the therapeutic effect of the act of touching. Therapeutic touch, alternatively known as healing touch, is a complementary/alternative treatment method applied by touching energy points in the body. Therefore, this study was planned to examine the effect of therapeutic touch applied to hemodialysis patients on perceived stress and comfort levels. This study, planned as a randomized experimental study with a pre-test-post-test intervention control group, will be a study on dialysis patients receiving treatment at the hemodialysis unit of Fırat University Hospital between June 2025-June 2026. The sample will consist of a minimum of 60 dialysis patients (30 intervention, 30 control) who meet the research criteria and accept the study. The patients in the intervention and control groups will first be informed about the application before starting the application and their verbal and written consents will be obtained. Then, the Patient Identification Form, Visual Analog Scale-Comfort (VAS-Comfort), Hemodialysis Comfort Scale (HKS) and Perceived Stress Scale (PSS) will be applied and the 1st measurement will be obtained. The application will last approximately 15-30 minutes for the patients in the intervention group every three days. After three days of alternate application, data forms will be filled in again for patients and 2nd measurements will be obtained. During this period, no intervention will be made to patients in the control group and only the normal treatment protocol will be applied. At the end of three days, data forms will be filled in again and 2nd measurements will be obtained. In the analysis of data; frequency and percentage analyses, chi-square analysis, standard deviation, t-test in dependent groups, t-test analysis in independent groups will be performed.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months of hemodialysis treatment • Cognitive function is in place

Exclusion Criteria:

* Those with communication problems
* Those who do not agree to participate in the study
* Patients who receive traditional treatment for the disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale - Comfort | At the end of the third day
  The Visual Analog Scale was developed by Price et al. (1983) to assess pain intensity. In previous studies, VAS was also used to determine the comfort levels of patients. In this study, VAS was used to assess the comfort levels of patients. A score of 0 on the scale for comfort assessment indicates "I have no comfort at all", and a score of 10 indicates "I have great comfort".
Hemodialysis Comfort Scale | At the end of the third day
  The scale, developed by Şahin Orak and colleagues (2017) to determine the comfort levels of hemodialysis patients, consists of 9 items and two sub-dimensions. The responses to item 4 of the scale are scored as "never" 1 point, "very rarely" 2 points, "sometimes" 3 points, "very often" 4 points and "always" 5 points. The scores given to the other items (1-3, 5-9) are scored in reverse: "never" 5 points, "very rarely" 4 points, "sometimes" 3 points, "very often" 2 points and "always" 1 point. The scale has two sub-dimensions: "Relaxation" (items 7-9) and "Overcoming" (items 1-6). The total score evaluation of the scale and its sub-dimensions is determined by calculating the average score. The increase in the total score obtained from the scale indicates that the comfort level increases. In the validity and reliability study of the developed scale, the Cronbach alpha value for the total scale was determined as 0.87.
Perceived Stress Scale | At the end of the third day
  The Perceived Stress Scale was developed by Cohen et al. in 1983 to determine the level of stress that threatens human health. Its Turkish validity and reliability were determined by Eskin et al. (2013). The scale consists of 2 factors: "insufficient self-efficacy" and "stress" perception. The scale is a 5-point Likert-type scale and consists of 14 items. As the scores obtained from the scale increase, the stress level perceived by the person also increases. PSS scores range from 0 to 56, with a score range of 0-35 indicating a normal stress level and a score range of 35-56 indicating that the individual is under stress. In the original study of the scale, the Cronbach Alpha coefficient was found to be 0.84

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat university, Elâzığ, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No